CLINICAL TRIAL: NCT03174171
Title: Open-label Study on Treatment of Primary Aldosteronism With Everolimus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPA
Record Dates: First submitted 2017-05-24; First posted 2017-06-02 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Primary Aldosteronism
Keywords: Everolimus, mTor inhibitor
MeSH Terms: conditions — Hyperaldosteronism | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Everolimus 0.75 mg b.i.d. orally for 14 days.
  Interventions: Drug: Everolimus 0.75 mg

INTERVENTIONS:
Drug: Everolimus 0.75 mg — Everolimus 0.75 mg b.i.d. orally for 14 days.

SUMMARY:
The overall objective is to evaluate everolimus as an aldosterone-lowering drug in the treatment of primary hyperaldosteronism.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate everolimus as an aldosterone-lowering drug in treatment of primary aldosteronism.

Primary aldosteronism is defined as a group of disorders in which aldosterone production is inappropriately high and relatively autonomous from regulation by the renin-angiotensin-aldosterone system. It often presents with increased blood pressure and constitutes the most common cause of endocrine hypertension. It is associated with an increased risk of cardiovascular complications, structural and functional renal abnormalities and metabolic syndrome. The goal of primary aldosteronism treatment is to prevent mortality and morbidity associated with hypertension, hypokalemia and direct aldosterone-associated organ damage.

Treatment depends on the underlying cause of primary aldosteronism. In general, patients with aldosterone-producing adenoma and unilateral adrenal hyperplasia are recommended to have adrenalectomy while patients with bilateral adrenal hyperplasia and those not willing to obtain surgery are offered targeted treatment with mineralocorticoid receptor antagonists. However, the use of mineralocorticoid receptor antagonist is related to side effects that include breast tenderness, gynecomastia, sexual dysfunction and menstrual irregularities.

The primary purpose of this proof-of-concept study is to evaluate whether inhibition of adrenocortical mammilian target of rapamycin (mTOR) signalling with everolimus decreases circulating aldosterone levels. The study also aims to determine whether potential changes in aldosterone levels result solely from a direct effect of everolimus on the adrenal gland or could be caused by changes in aldosterone metabolism and/or levels of canonical regulators of adrenal function (ACTH, AngII). The secondary purpose of this study is to test whether everolimus treatment ameliorates hypertension, improves cardiac function and to better understand molecular mechanisms leading to the development of primary aldosteronism.

Participants will receive Everolimus 0.75mg b.i.d. orally for a duration of 14 days. Blood pressure measurements, haemodynamic measurements, blood tests, 24h urine collection and saline Infusion tests will be conducted in order to compare changes in blood pressure, cardiac and kidney function, aldosterone and steroid hormone metabolite levels, activity of the renin-angiotensin-aldosterone system before and after treatment.

In patients undergoing adrenalectomy, adrenocortical cells will be isolated and primary adrenocortical cell cultures will be established from excised adrenal glands. Cultured cells will be treated with mTOR inhibitors and their proliferation and steroidogenic potential will be assessed. Cells treated with mTOR inhibitors will be subjected to transcriptomic, proteomic and phosphoproteomic analyses that will allow identification of mTOR signaling effectors in the adrenal cortex and to better understand molecular mechanisms leading to the development of primary aldosteronism.

ELIGIBILITY:
Inclusion Criteria:

* Patient with primary aldosteronism
* Age ≥ 18 years
* Office blood pressure <160/90 mmHg on antihypertensive therapy
* For subjects with reproductive potential, willingness to use contraceptive measures adequate to prevent the subject or the subject's partner from becoming pregnant during the study

Exclusion Criteria:

* Signs of current infection
* Neutropenia (leukocyte count < 1.5 × 109/L or absolute neutrophil count (ANC) < 0.5 × 109/L)
* Anemia (hemoglobin < 11 g/dL for males, < 10 g/dL for females)
* Clinically significant kidney or liver disease (creatinine > 1.5 mg/dL, aspartate aminotransferase (AST)/alanine aminotransferase (ALT) > 2 × ULN, alkaline phosphatase > 2 × ULN, total bilirubin > 1.5 × ULN)
* Current immunosuppressive treatment or documented immunodeficiency
* Uncontrolled congestive heart failure
* Currently pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2018-06-25 (Actual)

PRIMARY OUTCOMES:
Aldosterone level | 28 days
  Change in aldosterone level after saline infusion test after the treatment period (Day 15) and after the washout period (Day 28) compared to baseline (Day 0).

SECONDARY OUTCOMES:
Blood pressure values | 28 days
  Change in mean systolic and diastolic blood pressure during standardized office and home blood pressure measurement after the treatment period (Day 15) and after the washout period (Day 28) compared to baseline (Day 0).
Kidney function | 28 days
  Change in albumin in 24 hour-urine after the treatment period (Day 15) and after the washout period (Day 28) compared to baseline (Day 0).
Steroid hormones in serum | 28 days
  Change in steroid hormones in serum in 24h-urine after the treatment period (Day 15) and after the washout period (Day 28) compared to baseline (Day 0).
Level of plasma renin activity | 28 days
  Change in Renin-angiotensin-aldosterone System after the treatment period (Day 15) and after the washout period (Day 28) compared to baseline (Day 0).
Level of Potassium | 28 days
  Change in potassium level and need of potassium substitution after the treatment period (Day 15) and after the washout period (Day 28) compared to baseline (Day 0).
Steroid hormone metabolites in urine | 28 days
  Change in steroid hormone metabolites in 24h-urine after the treatment period (Day 15) and after the washout period (Day 28) compared to baseline (Day 0).
Level of plasma ACTH | 28 days
  Change in the Renin-angiotensin-aldosterone system after the treatment period (Day 15) and after the washout period (Day 28) compared to baseline (Day 0).
Level of plasma angiotensin II (ATII) | 28 days
  Change in the Renin-angiotensin-aldosterone system after the treatment period (Day 15) and after the washout period (Day 28) compared to baseline (Day 0).

CONTACTS AND LOCATIONS:
Overall Officials: Marc Y Donath, Prof., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No